CLINICAL TRIAL: NCT03717818
Title: Mechanisms of Change in Brief Treatment for Borderline Personality Disorder: A Randomized Controlled Trial
Brief Title: Mechanisms of Change in Brief Treatment for Borderline Personality Disorder
Acronym: BPDCHANGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Ueli Kramer, PD Dr. phil. Head of Research, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-02167
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Good Psychiatric Management-Brief (Experimental)
  Interventions: Behavioral: Good Psychiatric Management - Brief
- Treatment as Usual-Brief (Placebo Comparator)
  Interventions: Behavioral: treatment as usual

INTERVENTIONS:
Behavioral: Good Psychiatric Management - Brief — specific interventions as defined by Gunderson and Links (2014)
  Arms: Good Psychiatric Management-Brief
Behavioral: treatment as usual — non-specific intervention
  Arms: Treatment as Usual-Brief

SUMMARY:
The present two-arm randomized controlled study aims at testing the effects (i.e., symptom reduction) and the underlying mechanisms of change associated with a brief psychiatric treatment (10 sessions over 4 months), compared with treatment as usual. Participants undergo assessments at four points (intake, 2 months, discharge and 12 month follow-up). In addition to symptom measures, all individuals undergo a two-step assessment for the potential mechanisms of change (i.e., emotion and socio-cognitive processing): a) behavioural and b) neurofunctional. We hypothesize that change in the mechanisms explains the treatment effects. The present study uses an innovative treatment of BPD and at the same time a sophisticated assessment procedure to demonstrate the critical role of psychobiological change in emotion and sociocognitive processing in brief treatments. It will help increase the effectiveness of initial treatment phase for BPD and help diminish the societal burden of disease related with BPD. This study is funded by the Swiss National Science Foundation (SNSF).

ELIGIBILITY:
Inclusion Criteria:

* Borderline Personality Disorder
* age between 18 and 35

Exclusion Criteria:

* non-mastery in French
* neurological disorders
* schizophrenia (according to DSM-5)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
ZAN-BPD (Zanarini Borderline Personality Disorder Scale; Zanarini, 2003) | 4 months
  measures borderline symptomatology from an dimensional perspective, ranges between 0 and 36 (36 being the most symptomatic), global score (sum of all 9 items coded between 0 and 4) used.

SECONDARY OUTCOMES:
OQ-45 (Outcome Questionnaire-45.2, Lambert et al., 2004) | 4 months
  measures the level of problems (distress, social and interpersonal) on a scale ranging from 0 to 180 (45 items coded between 0 and 4, 4 being the most symptomatic). A total sum score will be used
BSL-23 (Borderline Symptom List, Short Version; Bohus et al., 2009) | 4 months
  measures the intensity of borderline symptoms using a mean score of the 23 items ranging between 0 and 4 (4 being the most symptomatic), the mean score will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry-CHUV, University of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Kramer U, Kolly S, Maillard P, Pascual-Leone A, Samson AC, Schmitt R, Bernini A, Allenbach G, Charbon P, de Roten Y, Conus P, Despland JN, Draganski B. Change in Emotional and Theory of Mind Processing in Borderline Personality Disorder: A Pilot Study. J Nerv Ment Dis. 2018 Dec;206(12):935-943. doi: 10.1097/NMD.0000000000000905. PMID 30507735
- [Derived] Kramer U, Grandjean L, Machinea JB, Beuchat H, Ranjbar S, de Roten Y, Despland JN, Conus P, Kolly S. Emotional processing as mechanism of change in brief good psychiatric management for borderline personality disorder: results of a randomized controlled trial. BMC Psychiatry. 2024 Dec 18;24(1):921. doi: 10.1186/s12888-024-06370-2. PMID 39696018
- [Derived] Kramer U, Grandjean L, Beuchat H, Kolly S, Conus P, de Roten Y, Draganski B, Despland JN. Mechanisms of change in brief treatments for borderline personality disorder: a protocol of a randomized controlled trial. Trials. 2020 Apr 16;21(1):335. doi: 10.1186/s13063-020-4229-z. PMID 32299512